CLINICAL TRIAL: NCT06933719
Title: Research Into Perinatal Care, Its Complications and Exposure to Multiple Factors (PRECEE2)
Brief Title: PRECEE2 Perinatal Research
Acronym: PRECEE2
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/688
Record Dates: First submitted 2025-03-27; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Study on existing health data — Study on existing health data

SUMMARY:
The aim of this study is to analyze the relationship between complications and adverse pregnancy outcomes and exposure to environmental factors in women living in Franche-Comté who gave birth between 2011 and 2025 at Besancon University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Women who gave birth at the CHUB between 01/01/2011 and 12/31/2025
* who have not expressed any objection to the processing of their data.

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Subject is within the exclusion period of another study or is excluded from the "national volunteer file".
* Subject refusing the collection of his/her medical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who gave birth at the CHUB between 01/01/2011 and 12/31/2025
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
pregnancy complications | at birth
  Description of Pregnancy Complications

IPD SHARING:
Plan to Share IPD: Undecided